CLINICAL TRIAL: NCT02883010
Title: A Randomised Controlled Study to Compare Surgical Site Complication Incidence in Subjects Receiving PICO or Standard Care Following Colorectal Surgery
Brief Title: Comparison of Surgical Incision Complications in Patients Receiving PICO or Standard Care Following Colorectal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT1602PIC
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Wounds and Injuries
Keywords: Surgical incision; surgical complication; NPWT; negative pressure; colorectal surgery; dehisced
MeSH Terms: conditions — Wounds and Injuries; Surgical Wound | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICO (Experimental): Single use NPWT (PICO Softport V1.6)
  Interventions: Device: PICO Softport V1.6
- Standard care (Other): Gauze dressing, Film dressing, foam dressing, skin glue, no dressing
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: PICO Softport V1.6 — PICO is a Single-Use Negative Pressure Wound Therapy (NPWT) System consisting of a small portable pump, 2 lithium batteries, 2 dressings and fixation strips. The system is capable of delivering up to 80 mm Hg negative pressure to a wound or surgical incision site and managing low to moderate levels of exudate or fluid generated by the wound or incision. The therapy may be administered for up to 2 weeks.
  Arms: PICO
Other: Standard Care — Care path normally used by the hospital
  Arms: Standard care

SUMMARY:
Surgical Site Complications (SSC's) are responsible for increased morbidity in patients undergoing surgery resulting in prolonged length of stay in the hospital while increasing treatment and hospital costs dramatically. Negative Pressure Wound Therapy (NPWT) use on closed incisions has been reported in the literature to reduce SSC's including Surgical Site Infections (SSI's), with many promising studies in general surgery, including some studies using single use NPWT. However, to date, there are very few randomised controlled trials (RCT's) using this intervention. When using PICOTM (NPWT) for this indication, patients may be discharged from hospital earlier, with the negative pressure incision management in place. This has implications in terms of cost savings for the health care system and enables the patient to be able to return to their normal daily routine more quickly. The hypothesis of this study is that PICO NPWT will reduce frequency of SSC's, in a 30 day follow up period, as compared to standard care in patients undergoing colorectal procedures.

ELIGIBILITY:
INCLUSION CRITERIA

1. The subject or legal guardian must provide written informed consent (reference section 9.1).
2. Subjects eighteen (18) years of age or older.
3. Willing and able to make all required study visits.
4. Able to follow instructions.
5. Males or females.
6. Subject must be classified as a high risk patient in terms of likelihood for SSC's (i.e., heavy smoker (more than 20 cigarettes per day), diabetic, BMI ≥ 30, immunocompromised) or be treated as an emergency patient with obstructed bowel, perforated bowel or peritonitis and be undergoing any of the following procedures:- Left hemicolectomy, right hemicolectomy, extended right hemicolectomy, sigmoidectomy, anterior rectum resection, total colectomy.

EXCLUSION CRITERIA

1. Contraindications or hypersensitivity to the use of the investigational product or its components (e.g., silicone adhesives and polyurethane films [direct contact with incision], acrylic adhesives [direct contact with skin], polyethylene fabrics and super-absorbent powders [polyacrylates]) within the dressing.
2. Subjects with extremely fragile skin who require the use of SECURA non-sting barrier skin wipes and have hypersensitivity to the ingredients in the wipes.
3. Participation in another clinical trial (with use of investigational medicinal product or medical device) within thirty (30) days of Visit 1 or during the study.
4. Subjects with skin features (e.g., tattoos, pre-existing scarring) which, in the opinion of the Investigator, could interfere with the study assessments.
5. Subjects who have participated previously in this clinical trial.
6. Subjects with a reference incision (that is the largest incision that is made during the surgery and the one that is allocated to study treatment) less than 8cm.
7. Subjects with incisions exceeding 40 cm in length.
8. Subjects with incisions that are actively bleeding unless homeostasis has been achieved (to be confirmed during surgery).
9. Patients attending for a re-operation within the last 3 months.
10. Patients undergoing a procedure as part of palliative care (to be confirmed during surgery).
11. Patients with a systemic infection (that is not related to perforated bowel or peritonitis) at the time of surgery.
12. Patients with a known history of poor compliance with medical treatment.
13. Patients who also have a gynaecological procedure carried out during the colorectal procedure.
14. Patients other than those with a disease known to affect the immune system that are on steroids or other immune modulators known to impact healing.
15. Patients with a genetic or acquired healing defect.
16. Exposure of blood vessels, organs, bone or tendon within the incision (to be confirmed during surgery).
17. Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of complications in each group | 30 days

SECONDARY OUTCOMES:
Dehiscence incidence during a 30-day follow-up period | 30 days
Haematoma incidence during a 30-day follow-up period | 30 days
Seroma incidence during a 30-day follow-up | 30 days
Time to surgical incision closure | 30 days
Total length of hospital stay, including readmissions during a 30-day follow-up period | 30 days
Time to initial discharge during a 30-day follow-up period | 30 days
Total number of readmissions during a 30-day follow-up period | 30 days
To compare PICO against Standard Care for differences in Health Related Quality of Life (HRQoL) using SF-12 over the 14-day and 30-day follow-up period | 30 days
Overall per subject treatment cost for PICO and Standard Care | 30 days
Cost per Quality Adjusted Life Year (QALY) within a 30-day follow-up period | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Beate Hanson, MD, PhD, Study Chair — Vice President, Global Clinical Strategy

IPD SHARING:
Plan to Share IPD: No